CLINICAL TRIAL: NCT06210165
Title: Effects of Sugammadex and Conventional Reversal on Lung Function in Laparoscopic Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhendra Hardy Mohamad Zaini (Other)
Responsible Party: Sponsor-Investigator, Rhendra Hardy Mohamad Zaini, Associate Professor, Dr, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: USM/JEPeM/22050289
Record Dates: First submitted 2023-09-27; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Atelectasis, Postoperative; Pulmonary Function; Newborn, Abnormal
MeSH Terms: conditions — Pulmonary Atelectasis; Antisocial Personality Disorder | interventions — Sugammadex; Neostigmine; Atropine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex (Experimental): IV Sugammadex 4mg/kg once after Train of Four ratio 0.7 to 0.9
  Interventions: Drug: Sugammadex
- Neostigmine and atropine (Active Comparator): IV Neostigmine 40mcg/kg and IV Atropine 10mcg/kg once after Train of Four ratio 0.7 to 0.9
  Interventions: Drug: Neostigmine and atropine

INTERVENTIONS:
Drug: Sugammadex — IV Sugammadex 4mg/kg stat once TOF ratio 0.7-0.9 after completing surgery
  Other Names: Interventional Reversal
  Arms: Sugammadex
Drug: Neostigmine and atropine — IV neostigmine 40mcg/kg in combination with IV atropine 10mcg/kg stat once TOF ratio 0.7-0.9 after completing surgery
  Other Names: Conventional reversal
  Arms: Neostigmine and atropine

SUMMARY:
The goal of this clincal trial is to determine the differences in few parameter of lung function (ie Forced Vital Capacity (FCV)) between Sugammadex and conventional reversal in laparoscopic abdominal surgery. The main questions it aims to answer are:

1. Is there differences in the pulmonary function test preoperative and post extubation between Sugammadex and conventional reversal in laparoscopic abdominal surgery?
2. Is there differences in the size of atelectasis area between Sugammadex and conventional reversal in laparoscopic abdominal surgery?
3. Is there differences between sugammadex and conventional reversal in postoperative mean length of stay in laparoscopic abdominal surgery?

Participants will be asked

1. to do baseline spirometry before operation
2. to be examined for lung ultrasound before operation
3. to be given either sugammadex or neostigmine as reversal after operation is completed
4. to repeat spirometry after operation for few times
5. to be examined for lung ultrasound after operation

Researcher will compare sugammadex group and conventional group to see if any difference in term of lung function, size of atelectasis and length of stay.

DETAILED DESCRIPTION:
Postoperative Pulmonary Complications (PPCs) are not uncommon. They increase healthcare resource usage as well as increase mortality of the patients. There are many definitions published in literature which can be considered as a composite outcome measure. This includes atelectasis, respiratory infection, respiratory failure, pleural effusion, pneumothorax, bronchospasm as well as aspiration pneumonitis (Jammer et al., 2015). After induction of general anaesthesia, the respiratory system changes occur immediately: muscle function and respiratory drive change, volume of lungs decreases, and atelectasis occurs in more than 75% of patients who were given neuromuscular blocking agent,

The problem and rationale of the study are described in the following paragraphs according to three postoperative conditions, 1) pulmonary function, 2) atelectasis, and 3) postoperative length of stay:

Postoperative pulmonary complications are one of the major problems after a surgery. Even if the surgery was successful, patient will still be facing morbidity or even mortality after the surgery. The risk of PPCs increases in patients having respiratory problem such as asthma, chronic obstructive pulmonary disease (COPD) and smoker . Many studies have shown the comparison between Sugammadex and conventionally used Neostigmine with respect to PPCs. However, studies regarding Sugammadex and Neostigmine in term of pulmonary function postoperative are still scarce as only two studies were found to comment directly on pulmonary function by using spirometry between neostigmine and sugammadex. In those studies, it shown that no significant different in term of spirometry volume postoperative between sugammadex and neostigmine . The authors believed postoperative analgesia plays important role in reported preservation of FVC.

Atelectasis as one of the commonest PPC can be worsen especially in laparoscopic surgery by the effect of Trendelenburg position and pneumoperitoneum. Residual paralysis even not in such condition (Trendelenburg, pneumoperitoneum) has been demonstrated to contribute to impaired upper airway and pulmonary function as well as respiratory adverse events in PACU and might make the atelectasis even worse. This shows that there is a need for an effective and complete reversal of neuromuscular blocker to prevent such event.

The length of stay after operation is important as it may present the quality of the health care system. However, there are many factors that can contribute to length of stay postoperative where postoperative pulmonary complications is one of the greatest contributors. A study which conducted by Ledowski et al. on elderly group more than 75 years old in centres across 5 countries (South Korea, Malaysia, Australia, Hungary, Netherlands) regarding comparison neostigmine and sugammadex showed that there is no significant different in length of stay. Only in Malaysia Ledowski et.al found that there is significant difference in terms of length of stay. Thus, further study is needed to compare the post operative length of stay between patients reversed with Sugammadex and Neostigmine.

From reviews of literatures, there is a gap in studies involving comparison of the effect of sugammadex and neostigmine as reversal. The gap lies in 1) the scarcity of studies involving Sugammadex and Neostigmine in terms of pulmonary function postoperative, 2) a need for an effective and complete reversal of neuromuscular blocker, and 3) further study on postoperative length of stay is needed.

Research Question(s)

1. Are there differences in the pulmonary function test preoperative and post extubation between Sugammadex and conventional reversal in laparoscopic abdominal surgery?
2. Are there differences in the size of atelectasis area between Sugammadex and conventional reversal in laparoscopic abdominal surgery?
3. Are there differences between sugammadex and conventional reversal in postoperative mean length of stay in laparoscopic abdominal surgery?

Thus, we formulate from the research questions with null hypothesis as below:

1. There is no difference in Forced Vital Capacity (FVC), Forced Expiratory Volume in the first second (FEV1), and FEV1/FVC preoperative and post extubation between Sugammadex and conventional reversal group in laparoscopic abdominal surgery
2. There is no difference in the size of atelectasis area using ultrasonography preoperative and post extubation between sugammadex and conventional reversal in laparoscopic abdominal surgery
3. There is no difference in mean postoperative length of stay (days) in hospital between sugammadex and conventional reversal in laparoscopic abdominal surgery Objective General: To compare the effect on lung function between sugammadex and conventional reversal in laparoscopic abdominal surgery

Specific:

1. To compare the Forced Vital Capacity (FVC), Forced Expiratory Volume in the first second (FEV1), and FEV1/FVC using portable spirometry preoperative and post extubation between sugammadex and conventional reversal in laparoscopic abdominal surgery
2. To identify and compare the size of atelectasis area using ultrasonography preoperative and post extubation between sugammadex and conventional reversal in laparoscopic abdominal surgery
3. To compare mean postoperative length of stay (days) in hospital between sugammadex and conventional reversal in laparoscopic abdominal surgery

All data collection will be collected at Hospital Universiti Sains Malaysia, Kubang Kerian. Patient will be identified based on inclusion and exclusion criteria from locations listed below:

1. Anaesthesia clinic
2. In the ward, during review by preanaesthesia review for the elective operation in the following day
3. In the ward, when cases are notified for operations as emergency case
4. In operation theatre, when cases notified arrived for emergency operation.

The informed consent will be obtained from patients either in ward, clinics or in Operation Theatre during emergency premedication at the airlock. The patient will be given ample time to decide on the participation. The consent for general anaesthesia also will be taken as part of standard practice. Related information such as fasting hours will be conveyed.

After consent is explained and taken, baseline spirometry and lung ultrasound (LUS) will be performed before general anaesthesia given, either in wards, clinics or operation theatre. This to get the baseline of pulmonary function as well as lung images. Spirometry will be performed following international recommendations but with patients in a semi recumbent position (40 degree) as recommended for postoperative position (Graham et al., 2019). FVC, FEV1 and forced expiratory flow 25-75% will be measured and recorded. Changes in lung aeration will be studied by LUS with the patient in the same position. LUS will be conducted on each lung in sagittal section at three predefined areas: parasternal, medial axillary line, and posterior axillary line (Lichtenstein, 2014). Brightness will be adjusted in setting to the brightest level in the bony surface of ribs. After that, the scale in cm2 will be set according to image resolutions in pixels. Presence of hepatization pattern of lung tissue will indicate the collapsed area. This suggesting atelectasis is present. The area will be measured in each area by taking the longest length vertically and horizontally, during end-expiration after freezing the image. The sum of all six area will be added, recorded and considered as size of atelectasis.

Patient will be induced by anaesthesiologist in-charge as routine clinical practice. Neuromuscular block will be performed using rocuronium prior intubation and monitored by train-of-four (TOF) Watch. Anaesthesiologist will be allowed to maintain TOF level according to usual criteria. Desflurane or sevoflurane will be used as maintenance.

After operation is completed, patient will be randomly assigned to receive either sugammadex 4mg/kg or neostigmine 40mcg/kg in combination with atropine 10mcg/kg using sealed opaque envelopes. The reversal will be given once the TOF ratio ranging between 0.7 to 0.9 as the diaphragm muscles and tidal volume are already back to normal (Wardhana et al., 2019). An extra dose of reversal is permitted by protocol, when needed, at the discretion of the attending anaesthesiologist. Patient will be extubated as usual local practice and will be sent to postoperative recovery room.

In order to ensure patient able to obey command, new spirometry will be performed in the postoperative recovery room only after 20 minutes of extubation with the same procedure and position used in the preoperative determinations. Postoperative clinical management will be conducted according to clinical preferences and local protocol. Additional lung ultrasound scan is performed as well at 20 minutes post extubation, just after spirometry. The spirometry is repeated at 60 minutes post extubation. All measurements will be recorded.

Another spirometry will be done 24H after operation in ward in the same manner and measurement will be recorded. The patient will be followed up in ward until discharge and the length of stay postoperative will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed / suspected: appendicitis or cholelithiasis
* Planned for laparoscopic operation under general anaesthesia
* ASA I-III

Exclusion Criteria:

1. Unstable haemodynamic status
2. Patient refusal to participate
3. Altered mental status, cognitive function or mental disorder
4. Admission to postoperative care unit (PACU) under mechanical ventilation
5. Hypersensitivity to any of the drugs
6. Acute or chronic lung diseases
7. Neuromuscular disorders
8. Myocardial infarction or coronary occlusion three months prior surgery
9. Obesity BMI more or equal 30
10. Intubation prior operating room arrival
11. Pregnancy
12. Converted to open surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Lung Function | Preoperative (Hour 1)to 24H post extubation (Hour 24)
  compare the Forced Vital Capacity (FVC), Forced Expiratory Volume in the first second (FEV1), and FEV1/FVC using portable spirometry preoperative and post extubation between sugammadex and conventional reversal in laparoscopic abdominal surgery

SECONDARY OUTCOMES:
Atelectasis | Preoperative (baseline) and 20 minutes post extubation
  compare the size of atelectasis area using ultrasonography preoperative and post extubation between sugammadex and conventional reversal in laparoscopic abdominal surgery.
Length of stay | Through study completion, an average one week
  compare mean postoperative length of stay (days) in hospital between sugammadex and conventional reversal in laparoscopic abdominal surgery

CONTACTS AND LOCATIONS:
Overall Officials: NIK MUHAMMAD 'AIZAT 'ADROS, MBBS, Principal Investigator — Hospital Universiti Sains Malaysia
Locations (1):
- University of Science Malaysia Hospital, Kubang Kerian, Kelantan, Malaysia

REFERENCES:
- [Background] Abola RE, Romeiser J, Rizwan S, Lung B, Gupta R, Bennett-Guerrero E. A randomized-controlled trial of sugammadex versus neostigmine: impact on early postoperative strength. Can J Anaesth. 2020 Aug;67(8):959-969. doi: 10.1007/s12630-020-01695-4. Epub 2020 May 13. PMID 32405975
- [Background] Alday E, Munoz M, Planas A, Mata E, Alvarez C. Effects of neuromuscular block reversal with sugammadex versus neostigmine on postoperative respiratory outcomes after major abdominal surgery: a randomized-controlled trial. Can J Anaesth. 2019 Nov;66(11):1328-1337. doi: 10.1007/s12630-019-01419-3. Epub 2019 Jun 4. PMID 31165457
- [Background] Amorim P, Lagarto F, Gomes B, Esteves S, Bismarck J, Rodrigues N, Nogueira M. Neostigmine vs. sugammadex: observational cohort study comparing the quality of recovery using the Postoperative Quality Recovery Scale. Acta Anaesthesiol Scand. 2014 Oct;58(9):1101-10. doi: 10.1111/aas.12389. Epub 2014 Sep 1. PMID 25179550
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310
- [Background] Echeverry G, Polskin L, Tollinche LE, Seier K, Tan KS, McCormick PJ, Fischer GW, Grant FM. ROUTINE USE OF SUGAMMADEX DOES NOT SHORTEN PACU LENGTH OF STAY: A PROSPECTIVE DOUBLE-BLINDED RANDOMIZED CONTROLLED TRIAL. Perioper Care Oper Room Manag. 2021 Sep;24:100199. doi: 10.1016/j.pcorm.2021.100199. Epub 2021 Jul 16. PMID 34504958
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Hristovska AM, Duch P, Allingstrup M, Afshari A. Efficacy and safety of sugammadex versus neostigmine in reversing neuromuscular blockade in adults. Cochrane Database Syst Rev. 2017 Aug 14;8(8):CD012763. doi: 10.1002/14651858.CD012763. PMID 28806470
- [Background] Hyman EC, Brull SJ. Clarification: Current Status of Neuromuscular Reversal and Monitoring, Challenges and Opportunities. Anesthesiology. 2017 Oct;127(4):730. doi: 10.1097/ALN.0000000000001795. No abstract available. PMID 28926458
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Kheterpal S, Vaughn MT, Dubovoy TZ, Shah NJ, Bash LD, Colquhoun DA, Shanks AM, Mathis MR, Soto RG, Bardia A, Bartels K, McCormick PJ, Schonberger RB, Saager L. Sugammadex versus Neostigmine for Reversal of Neuromuscular Blockade and Postoperative Pulmonary Complications (STRONGER): A Multicenter Matched Cohort Analysis. Anesthesiology. 2020 Jun;132(6):1371-1381. doi: 10.1097/ALN.0000000000003256. PMID 32282427
- [Background] Kim HY. Statistical notes for clinical researchers: Chi-squared test and Fisher's exact test. Restor Dent Endod. 2017 May;42(2):152-155. doi: 10.5395/rde.2017.42.2.152. Epub 2017 Mar 30. No abstract available. PMID 28503482
- [Background] Ledowski T, Szabo-Maak Z, Loh PS, Turlach BA, Yang HS, de Boer HD, Asztalos L, Shariffuddin II, Chan L, Fulesdi B. Reversal of residual neuromuscular block with neostigmine or sugammadex and postoperative pulmonary complications: a prospective, randomised, double-blind trial in high-risk older patients. Br J Anaesth. 2021 Aug;127(2):316-323. doi: 10.1016/j.bja.2021.04.026. Epub 2021 Jun 12. PMID 34127252
- [Background] Li L, Jiang Y, Zhang W. Sugammadex for Fast-Track Surgery in Children Undergoing Cardiac Surgery: A Randomized Controlled Study. J Cardiothorac Vasc Anesth. 2021 May;35(5):1388-1392. doi: 10.1053/j.jvca.2020.08.069. Epub 2020 Sep 3. PMID 32962936
- [Background] Lichtenstein DA. Lung ultrasound in the critically ill. Ann Intensive Care. 2014 Jan 9;4(1):1. doi: 10.1186/2110-5820-4-1. PMID 24401163
- [Background] Mazo V, Sabate S, Canet J. How to optimize and use predictive models for postoperative pulmonary complications. Minerva Anestesiol. 2016 Mar;82(3):332-42. Epub 2015 May 20. PMID 25990430
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Mongodi S, De Luca D, Colombo A, Stella A, Santangelo E, Corradi F, Gargani L, Rovida S, Volpicelli G, Bouhemad B, Mojoli F. Quantitative Lung Ultrasound: Technical Aspects and Clinical Applications. Anesthesiology. 2021 Jun 1;134(6):949-965. doi: 10.1097/ALN.0000000000003757. PMID 33819339
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Naguib M, Brull SJ, Johnson KB. Conceptual and technical insights into the basis of neuromuscular monitoring. Anaesthesia. 2017 Jan;72 Suppl 1:16-37. doi: 10.1111/anae.13738. PMID 28044330
- [Background] Nguyen TK, Nguyen VL, Nguyen TG, Mai DH, Nguyen NQ, Vu TA, Le AN, Nguyen QH, Nguyen CT, Nguyen DT. Lung-protective mechanical ventilation for patients undergoing abdominal laparoscopic surgeries: a randomized controlled trial. BMC Anesthesiol. 2021 Mar 30;21(1):95. doi: 10.1186/s12871-021-01318-5. PMID 33784987
- [Background] Norton M, Xara D, Parente D, Barbosa M, Abelha FJ. Residual neuromuscular block as a risk factor for critical respiratory events in the post anesthesia care unit. Rev Esp Anestesiol Reanim. 2013 Apr;60(4):190-6. doi: 10.1016/j.redar.2012.12.011. Epub 2013 Feb 28. PMID 23453244
- [Background] O'Reilly-Shah VN, Wolf FA, Jabaley CS, Lynde GC. Using a worldwide in-app survey to explore sugammadex usage patterns: a prospective observational study. Br J Anaesth. 2017 Aug 1;119(2):333-335. doi: 10.1093/bja/aex171. No abstract available. PMID 28854547
- [Background] Rivero-Yeverino D. [Spirometry: basic concepts]. Rev Alerg Mex. 2019 Jan-Mar;66(1):76-84. doi: 10.29262/ram.v66i1.536. Spanish. PMID 31013409
- [Background] Touw HR, Schuitemaker AE, Daams F, van der Peet DL, Bronkhorst EM, Schober P, Boer C, Tuinman PR. Routine lung ultrasound to detect postoperative pulmonary complications following major abdominal surgery: a prospective observational feasibility study. Ultrasound J. 2019 Sep 16;11(1):20. doi: 10.1186/s13089-019-0135-6. PMID 31523784
- [Background] Wang JF, Zhao ZZ, Jiang ZY, Liu HX, Deng XM. Influence of sugammadex versus neostigmine for neuromuscular block reversal on the incidence of postoperative pulmonary complications: a meta-analysis of randomized controlled trials. Perioper Med (Lond). 2021 Sep 20;10(1):32. doi: 10.1186/s13741-021-00203-6. PMID 34538277
- [Background] Wardhana A, Kurniawaty J, Uyun Y. Optimised reversal without train-of-four monitoring versus reversal using quantitative train-of-four monitoring: An equivalence study. Indian J Anaesth. 2019 May;63(5):361-367. doi: 10.4103/ija.IJA_94_19. PMID 31142879
- [Background] Yu J, Park JY, Lee Y, Hwang JH, Kim YK. Sugammadex versus neostigmine on postoperative pulmonary complications after robot-assisted laparoscopic prostatectomy: a propensity score-matched analysis. J Anesth. 2021 Apr;35(2):262-269. doi: 10.1007/s00540-021-02910-2. Epub 2021 Mar 8. PMID 33683444